CLINICAL TRIAL: NCT01930175
Title: A Randomized, Partial-blind, Placebo-controlled Trial Evaluating the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of VAY736 in the Treatment of Patients With Pemphigus Vulgaris
Brief Title: Study of Efficacy and Safety of VAY736 in Patients With Pemphigus Vulgaris
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study recruitment was terminated in Dec-2015 for strategic reasons related to the development of the compound.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAY736X2203
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Pemphigus Vulgaris
Keywords: Pemphigus vulgaris; pemphigus; blistering disease
MeSH Terms: conditions — Pemphigus | interventions — ianalumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): single dose iv of Placebo
  Interventions: Drug: Placebo
- VAY736 3 mg/kg (Experimental): single dose iv of VAY736 at a dose of 3mg/kg
  Interventions: Drug: VAY736
- VAY736 10 mg/kg (Experimental): single dose iv of VAY736 at a dose of 10mg/kg initiated following a safety review of patients receiving VAY736 3 mg/kg or placebo.
  Interventions: Drug: VAY736

INTERVENTIONS:
Drug: VAY736
  Other Names: Ianalumab
  Arms: VAY736 10 mg/kg; VAY736 3 mg/kg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study evaluated the efficacy, safety and pharmacokinetics of VAY736 in the treatment of patients with pemphigus vulagaris (PV).

DETAILED DESCRIPTION:
This was a non-confirmatory, randomized, partial-blind, placebo-controlled trial evaluating the efficacy, safety and pharmacokinetics (PK) of VAY736 in the treatment of PV patients.

A total of 13 patients were enrolled and randomized into the study. Of these 13 patients,seven were randomized to the 3 mg/kg VAY736 group, two were randomized to the 10 mg/kg VAY736 group and four were randomized to the placebo group.In the placebo group, three out of the four patients consented to open-label VAY736 treatment and received 10 mg/kg VAY736 after Week 24 onwards. Thus, a total of 12 patients received VAY736, 7 patients received 3 mg/kg and 5 patients 10 mg/kg.

The Screening period consisted of a Screening Visit performed within 28 days prior to randomization to assess patient eligibility. Following Screening, patients underwent pre-dose procedures which included assessment of their PV by Pemphigus Disease Area Index (PDAI), Autoimmune Bullous Skin disease Intensity Score (ABSIS) and Investigator Global Assessment (IGA), and blood sampling for PK endpoints. Patients then received the study drug, which was administered over approximately a 2 hour period. The patients remained in the study center overnight post-infusion for observation and for measurement of safety parameters and PK samples approximately 24 h post-infusion (start of infusion: ±2 h). Patients were then discharged from the study site and returned as per the schedule. Patients were evaluated at Week 1, Week 2 and Week 3, then every 3 weeks through to Week 12, and every 4 weeks through to Week 24. At Week 24, the blind was broken to confirm treatment allocation. If a patient was on placebo, such patient completing the Week 24 visit and after unblinding had the option of receiving open label VAY736 10mg/kg.

Recruitment was paused in Mar-2015 and at the time 13 patients were enrolled. The study recruitment was then terminated in Dec-2015 for strategic reasons related to the development of the compound.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 20 to 70 years of age
* Confirmed diagnosis of pemphigus vulgaris
* Presence of mild to moderate pemphigus vulgaris
* Patients must weight between 40 kg and 150 kg inclusive
* on a stable dose of oral corticosteriod therapy (with or without azathioprine or mycophenolate)

Exclusion Criteria:

* Pregnant or nursing (lactating) women
* Women of child-bearing potential unless they are using a highly effective method of birth control during dosing and for 4 months following study treatment
* Recent previous treatment with photo therapy, biological therapy, steroids, immunosuppresive agents (unless washout period applied)
* Active or recent history of clinically significant infection
* use of rituximab within 1 year Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-12-18 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (2):
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Philadelphia, Pennsylvania
- Novartis Investigative Site, Vienna, Austria
- Novartis Investigative Site, Sofia, BGR, Bulgaria
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=695

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 13 participants were enrolled and randomized into the study from Austria (1 center); Bulgaria (1 center); Taiwan (1 center); USA (2 centers).
Pre-assignment Details: The study was planned to be conducted in approximately 32 patients. However, after enrolling 13 patients, the recruitment was terminated due to strategic reasons related to the development of the compound.
Period: Core Study
Arm/Group | VAY736 3 mg/kg | VAY736 10 mg/kg | Placebo
Started | 7 | 2 | 4
Safety Analysis Set (Patients that received study drug) | 7 | 2 | 4
Pharmacokinetics (PK) Analysis Set (Patients with at least one PK measurement and no major protocol deviations affecting PK) | 7 | 2 | 0 (Placebo patients were excluded from the PK analyses)
Completed | 7 | 1 | 3
Not Completed | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1
Period: Open Label VAY736 10 mg/kg at Week 24
Arm/Group | VAY736 3 mg/kg | VAY736 10 mg/kg | Placebo
Started | 0 (Only patients originally randomized to Placebo were allowed to enter this Period.) | 0 (Only patients originally randomized to Placebo were allowed to enter this Period.) | 3 (Only patients originally randomized to Placebo were allowed to enter this Period.)
Completed | 0 | 0 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VAY736 3 mg/kg | VAY736 10 mg/kg | Placebo | Total
Number analyzed (Participants) | 7 | 2 | 4 | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.6 (10.45) | 35.0 (8.49) | 56.0 (8.83) | 50.4 (11.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 2 | 5
  Male | 4 | 2 | 2 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 1 | 1 | 4
  Caucasian | 4 | 1 | 3 | 8
  Other | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Pemphigus Disease Area Index (PDAI) at Week 12
Description: PDAI is specific cutaneous and mucosal disease activity assessment performed by investigator based on evaluation of lesions in well-defined anatomical locations. The score weighted for the number and size of lesions with score of 0 (absent) to 10 given for skin (12 body locations), scalp and mucous membrane showing disease activity (erosions/blisters or new erythema). Damage, such as post inflammatory hyperpigmentation or erythema from resolving lesion, scored separately from the main score as absent (0) or present (1) for each body area or scalp resulting in a score of 0 to 12 or 0 to 1, respectively. Thus, PDAI ranged from 0 to 263, with 250 points representing disease activity (120 points for skin activity; 10 points for scalp activity; 120 points for mucosal activity) and 13 points representing disease damage.
Time Frame: Week 12
Population: All evaluable patients.
Measure: Mean (Standard Deviation); unit: Score on the scale
Arm/Group | VAY736 3 mg/kg | VAY736 10 mg/kg | Placebo
Number analyzed (Participants) | 7 | 2 | 3
Score on the scale | 5.90 (1.836) | 10.15 (8.273) | 22.07 (25.628)

2. Secondary Outcome: Autoimmune Skin Disease Intensity Score (ABSIS) at Baseline and Week 12.
Description: The ABSIS Score is a quality- and quantity-based score for cutaneous and oral mucosal lesions combining the extent of the affected body surface area (BSA), the quality of the skin lesions and oral involvement. The ABSIS score ranged from 0 to 206 with 150 points for skin involvement, 11 points for oral involvement and 45 points for subjective discomfort during eating and drinking. A reduction from baseline (or, a negative change from baseline) in ABSIS indicates improvement in patients.
Time Frame: Baseline, Week 12
Population: All evaluable patients.
Measure: Mean (Standard Deviation); unit: Score on the scale
Arm/Group | VAY736 3 mg/kg | VAY736 10 mg/kg | Placebo
Number analyzed (Participants) | 7 | 2 | 4
Score on the scale
  Baseline | 13.26 (7.621) | 16.38 (12.905) | 33.75 (21.620)
  Week 12: number analyzed (Participants) | 7 | 2 | 3
  Week 12 | 2.19 (3.465) | 5.55 (7.707) | 16.17 (25.838)

3. Secondary Outcome: Change From Baseline in Investigator Global Assessment (IGA) at Week 12
Description: The IGA score ranges from 0 to 4 and the decrease or reduction from baseline in IGA score indicates improvement in patients.
  IGA score scale:
  0=Clear, 1=Near Clear, 2=Mild, 3=Moderate, 4=Severe active disease
Time Frame: Baseline, Week 12
Population: All evaluable patients.
Measure: Mean (Standard Deviation); unit: Score on the scale
Arm/Group | VAY736 3 mg/kg | VAY736 10 mg/kg | Placebo
Number analyzed (Participants) | 7 | 2 | 3
Score on the scale | -1.4 (0.79) | -1.0 (0.00) | -0.7 (0.58)

4. Secondary Outcome: VAY736 Serum Concentration - AUCinf
Description: The area under the serum concentration-time curve from time zero to infinity [mass × time / volume]. The concentration of VAY736 was measured in the serum.
Time Frame: predose, 2, 24 hours and weeks 1, 2, 3, 6, 9, 12, 16, 20, 24 and approximately 52 weeks
Population: PK analysis set: Patients with at least one PK measurement and no major protocol deviations affecting PK
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | VAY736 3 mg/kg | VAY736 10 mg/kg | Placebo
Number analyzed (Participants) | 7 | 2 | 0
day*ug/mL | 440 (114) | 1480 (231) |

5. Secondary Outcome: VAY736 Serum Concentration - AUClast
Description: The area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration [mass × time / volume]. The concentration of VAY736 was measured in the serum.
Time Frame: predose, 2, 24 hours and weeks 1, 2, 3, 6, 9, 12, 16, 20, 24 and approximately 52 weeks
Population: PK analysis set: Patients with at least one PK measurement and no major protocol deviations affecting PK
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | VAY736 3 mg/kg | VAY736 10 mg/kg | Placebo
Number analyzed (Participants) | 7 | 2 | 0
day*ug/mL | 440 (114) | 1480 (231) |

6. Secondary Outcome: VAY736 Serum Concentration - Cmax
Description: The observed maximum serum concentration following drug administration [mass / volume]. The concentration of VAY736 was measured in the serum.
Time Frame: predose, 2, 24 hours and weeks 1, 2, 3, 6, 9, 12, 16, 20, 24 and approximately 52 weeks
Population: PK analysis set: Patients with at least one PK measurement and no major protocol deviations affecting PK
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | VAY736 3 mg/kg | VAY736 10 mg/kg | Placebo
Number analyzed (Participants) | 7 | 2 | 0
ug/mL | 77.1 (13.0) | 230 (2.83) |

7. Secondary Outcome: VAY736 Serum Concentration - Tmax
Description: Tmax is the time to reach the maximum concentration after drug administration [time]. The concentration of VAY736 was measured in the serum.
Time Frame: predose, 2, 24 hours and weeks 1, 2, 3, 6, 9, 12, 16, 20, 24 and approximately 52 weeks
Population: PK analysis set: Patients with at least one PK measurement and no major protocol deviations affecting PK
Measure: Median (Full Range); unit: Hours
Arm/Group | VAY736 3 mg/kg | VAY736 10 mg/kg | Placebo
Number analyzed (Participants) | 7 | 2 | 0
Hours | 2.05 [2.00 to 2.22] | 2.11 [2.00 to 2.22] |

8. Secondary Outcome: VAY736 Serum Concentration - T1/2
Description: T1/2 is the terminal elimination half-life [time]. The concentration of VAY736 was measured in the serum.
Time Frame: predose, 2, 24 hours and weeks 1, 2, 3, 6, 9, 12, 16, 20, 24 and approximately 52 weeks
Population: PK analysis set: Patients with at least one PK measurement and no major protocol deviations affecting PK
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | VAY736 3 mg/kg | VAY736 10 mg/kg | Placebo
Number analyzed (Participants) | 7 | 2 | 0
Days | 11.2 (2.01) | 15.4 (1.93) |

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study for up to 5 years.
Description: Any sign or symptom until end of study for up to 5 years.
Groups:
- Open Label VAY736 10 mg/kg: Patients randomized to placebo in period 1 received open label VAY736 10mg/kg at week 24.
Arm/Group | VAY736 3 mg/kg | VAY736 10 mg/kg | Placebo | Open Label VAY736 10 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/2 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/2 | 1/4 | 1/3
Other Adverse Events (participants affected / at risk) | 6/7 | 2/2 | 3/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VAY736 3 mg/kg (N=7) | VAY736 10 mg/kg (N=2) | Placebo (N=4) | Open Label VAY736 10 mg/kg (N=3)
Cataract (Eye disorders) | 0 | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pemphigus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VAY736 3 mg/kg (N=7) | VAY736 10 mg/kg (N=2) | Placebo (N=4) | Open Label VAY736 10 mg/kg (N=3)
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival recession (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Dermatophytosis of nail (Infections and infestations) | 1 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 1
Impetigo (Infections and infestations) | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 1
Oral fungal infection (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Amylase increased (Investigations) | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 1
Blood potassium increased (Investigations) | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT01930175/Prot_001.pdf
  • Statistical Analysis Plan (2017-07-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT01930175/SAP_000.pdf